CLINICAL TRIAL: NCT01123317
Title: Brain Blood Flow Changes Elicited by Oxytocin in Healthy and Schizophrenic Volunteers, an Assessment Using Positron Emission Tomography and 15-Oxygen Labeled Water
Brief Title: Brain Blood Flow Changes Elicited by Oxytocin in Volunteers With and Without Schizophrenia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Never started
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Robert Buchanan, Director, Maryland Psychiatric Research Center, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: HP-00041288
Record Dates: First submitted 2010-05-12; First posted 2010-05-14 (Estimated); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; PET; Oxytocin
MeSH Terms: conditions — Schizophrenia | interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oxytocin (Experimental): Subjects will be randomly assigned to either OT-Placebo or Placebo-OT order for PET scan drug administration and will receive the first of the two intranasal doses at Pet scan 1 and the second intranasal dose of the subsequent treatment at Pet Scan 2
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Subjects will be randomly assigned to either OT-Placebo or Placebo-OT order for PET scan drug administration and will receive the first of the two intranasal doses at Pet scan 1 and the second intranasal dose of the subsequent treatment at Pet Scan 2
  Other Names: Syntocinon

SUMMARY:
The purpose of this study is to assess how oxytocin delivered intranasally changes regional brain blood flow measured by positron emission tomography (PET) in conjunction with oxygen-15 labeled water in persons with schizophrenia. The objective is to better our understanding of oxytocin's role in the modulation of social judgment in schizophrenia and provide more information as to potential uses of oxytocin or a similar drug analog in treating certain features of schizophrenia and other neuropsychiatric disorders.

DETAILED DESCRIPTION:
Schizophrenia is a severely debilitating psychiatric disorder that afflicts approximately 1% of the population (American Psychiatric Association, 1994) and is a serious public health problem. The specific mechanism of schizophrenia remains unknown. Affective responsivity and adaptive social behaviors are fundamental impairments in people with schizophrenia. These features have a detrimental impact on function in many areas of daily life. Unfortunately, the brain mechanisms that underlie these problems are still not understood. This study will use positron emission tomography (PET) and regional cerebral blood flow (rCBF) measures to ascertain the timing (1.5 hour period) of OT action on absolute regional brain activity in schizophrenia (SZ) and healthy control (HC) subjects. Particular focus will be on the amygdala, ventral striatum, anterior hippocampus and hypothalamus (neural regions involved in affliative behavior). Subjects will be studied with intranasally administered oxytocin and placebo while at rest and while making judgments about emotional faces. This approach will tell us to what extent the amygdala and limbic system's physiological response to oxytocin is predictive of a subject's behavioral sensitivity to this neuropeptide. The elucidation of this information may have a significant impact on predicting functional outcome and novel drug treatments in schizophrenia.

Functional magnetic resonance imaging (MRI) studies show that oxytocin modulates the amygdala's response during social and emotional decisions. When administered intranasally, OT may be beneficial for the treatment of negative symptoms in schizophrenia by enhancing a person's affiliative behavior and diminishing distrust. It is not, however, known to what extent intranasal oxytocin modifies regional neurotransmission and human brain metabolism. There are at present no studies in animals or humans specifically examining the time course action of OT on whole brain activity.

ELIGIBILITY:
Inclusion Criteria:

* Normal volunteers: Age range: 18-55 years of age
* Normal Volunteers: No psychiatric illness in self; no psychotic illness in first degree relatives
* Normal Volunteers: No previous history of substance dependence in last 6 months; no substance abuse in last month
* Normal Volunteers: No contraindication for MRI scanning (i.e. cardiac pacemaker, prosthesis)
* Normal Volunteers: Not pregnant
* Normal Volunteers: No major medical illness (e.g. seizure disorder) or medication that affects brain structure (e.g. steroids)
* Normal Volunteers: Participation in Healthy Subject Recruitment protocol (HP-00042350).
* Patient Volunteers: DSM-IV diagnosis of schizophrenia
* Patient Volunteers: Voluntary and competent to sign an informed consent
* Patient Volunteers: No contraindication for MRI scanning (i.e. cardiac pacemaker, prosthesis)
* Patient Volunteers: No previous history of substance dependence in last 6 months; no substance abuse in last month
* Patient Volunteers: Not pregnant
* Patient Volunteers: No major medical illness other than schizophrenia that affects brain structure (e.g. seizure disorder); not currently taking medication other than that for schizophrenia that affects brain structure (e.g. steroids)
* Patient Volunteers: No diagnosis of Major Depressive Disorder within last 6 months
* Patient Volunteers: SANS Asociality global score 2 or greater
* Patient Volunteers: No change in antipsychotic medication (type and dose) within the last 4 weeks
* Patient volunteers: Age range: 18-55 years of age

Exclusion Criteria:

* Normal Volunteers: Age outside of specified range -Normal Volunteers: Psychiatric illness in self; psychotic illness in first- degree relative
* Normal Volunteers: Previous history of substance dependence in last 6 months; substance abuse in last month
* Normal Volunteers: Contraindication for MRI scanning (i.e. cardiac pacemaker, prosthesis)
* Normal Volunteers: Pregnant
* Normal Volunteers: Major medical illness (e.g. seizure disorder) or medication that affects brain structure (e.g. steroids)
* Patient Volunteers: Age outside of specified range
* Patient Volunteers: Contraindication for MRI scanning (i.e. cardiac pacemaker, prosthesis)
* Patient Volunteers: History of substance dependence in last 6 months; substance abuse in last month
* Patient Volunteers: Pregnancy
* Patient Volunteers: Major medical illness other than schizophrenia that affects brain structure; currently taking medication other than that for schizophrenia that affects brain structure
* Patient Volunteers: Diagnosis of Major Depressive Disorder within last 6 months
* Patient Volunteers: SANS Asociality global score < 2
* Patient Volunteers: Change in antipsychotic medication (type and dose) within the last 4 weeks

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-07; Primary Completion 2011-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Oxytocin induced rCBF changes | 2 years
  Oxytocin induced rCBF changes in the amygdala, ventral striatum, hypothalamus and anterior hippocampus (post-drug versus pre-drug, resting and task conditions

CONTACTS AND LOCATIONS:
Overall Officials: Henry Holcomb, M.D., Principal Investigator — MPRC
Locations (1):
- Maryland Psychiatric Research Center, Catonsville, Maryland, United States